CLINICAL TRIAL: NCT04415034
Title: Scalp Pruritus Measurement Using Visual Analog Scale and 5-d Itch Scale in Children With Pediculosis Capitis
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr. dr. Sandra Widaty, SpKK (K), Principal investigator, Indonesia University
Other Study IDs: 0920/UN2.F1/ETIK/2018
Record Dates: First submitted 2020-05-27; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Pediculus Capitis; Pruritus
Keywords: Pediculosis capitis; Scalp pruritus; VAS scale; 5-D itch scale; Quality of life
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediculosis capitis: Subjects with pediculosis capitis based on the findings of eggs, larva, or an adult parasite on the scalp or in the hair
  Interventions: Other: VAS and 5-D itch pruritus assessment

INTERVENTIONS:
Other: VAS and 5-D itch pruritus assessment — All subjects were evaluated for presence of pruritus using VAS and 5-D itch scale

SUMMARY:
Pediculosis capitis is a parasitic infestation that can cause scalp pruritus and quality of life disturbances. There are two objective measurement for pruritus, visual analog scale (VAS) and 5-D itch scale, which can assess the severity of the scalp pruritus and the latter can also asses the quality of life affected by pruritus. Even though VAS can not be used to evaluate the impact of pruritus on quality of life, it is very easy to use while 5-D itch scale is complex and not child-friendly.

The aim of this study is to determine the relationship between two different pruritus scales and to establish validity of pruritus VAS scale in evaluating quality of life in children with pediculosis capitis. We compare two pruritus scale on students with pediculosis of two boarding school in Bogor, West Java, Indonesia.

DETAILED DESCRIPTION:
This study used cross sectional design study.

Subjects with eligible criteria were included and informed consent from the parents or legal guardian were obtained.

The diagnosis of pediculosis capitis was made based on the findings of eggs, larva, or an adult parasite on the scalp or in the hair of the students. All subjects were asked for both VAS and 5-D itch scale.The VAS is categorized into five groups based on the point, as follows: 0 for no pruritus, <3 for mild pruritus, ≥ 3 - <7 for moderate pruritus, ≥ 7 - <9 for severe pruritus, and ≥ 9 for very severe pruritus. The 5-D itch scale consists of five parameters: duration, degree, direction, disability (sleep, leisure/social activities, housework/errands, work/school), and distribution of the pruritus with points ranging from one to five.

Data were recorded for statistical analysis, a chi-square test was used to determine the relationship between two categorical variables. The correlation coefficient between the VAS and 5-D itch scale was calculated using Spearman's rank correlation

ELIGIBILITY:
Inclusion Criteria:

* Students studying in Junior high school at Boarding School in Bogor with medium length hair who were clinically diagnosed with pediculosis capitis
* Willingness to participate as a research subject (to be interviewed and undergo physical examination), and after being explained the details of the study, granted the headmaster permission to sign consent in their name (informed assent)

Exclusion Criteria:

* Chemical treatment of PC within 10 days before the trial
* History of permethrin hypersensitivity
* Unwillingness to participate as a research subject
* Mild-to-severe secondary infection
* Long or short hair

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Female students
Study Population: Subjects with pediculosis capitis
Sampling Method: Non-Probability Sample
Enrollment: 357 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Pruritus severity (1) | Baseline, during examination
  Pruritus severity evaluated by visual analog scale (VAS)
Pruritus severity (2) | Baseline, during examination
  Pruritus severity evaluated by 5-D itch scale

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Widaty, MD, PhD, Principal Investigator — Department of Dermatology and Venereology, Faculty of Medicine Universitas Indonesia
Locations (1):
- Pesantren Al Hidayah Cibinong, Bogor, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided